CLINICAL TRIAL: NCT02061059
Title: Improving the Cost-effectiveness of Therapeutic Shoes for Diabetic Patients With a Previous Foot Ulcer Using an In-shoe Pressure Device
Brief Title: Cost-effectiveness of In-shoe Pressure Measurement for Therapeutic Shoes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-1-112.3
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus; Polyneuropathies
MeSH Terms: conditions — Diabetes Mellitus; Polyneuropathies | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- group 1 (Other): group is assigned to "block 1": shoemaker 1 produces shoes according to standard methods, shoemaker 2 uses plantar pressure measurements.
  group is assigned to "standard": wears shoes produced with standard procedure
  Interventions: Other: block 1; Other: standard
- group 2 (Other): group is assigned to "block 1": shoemaker 1 produces shoes according to standard methods, shoemaker 2 uses plantar pressure measurements
  group is assigned to "with measurements": wears shoes produced with plantar pressure measurements
  Interventions: Other: block 1; Other: with measurements
- group 3 (Other): group is assigned to "block 2": shoemaker 2 produces shoes according to standard methods, shoemaker 1 uses plantar pressure measurements
  group is assigned to "standard": wears shoes produced with standard procedure
  Interventions: Other: block 2; Other: standard
- group 4 (Other): group assigned to "block 2": shoemaker 2 produces shoes according to standard methods, shoemaker 1 uses plantar pressure measurements
  group is assigned to "with measurements": wears shoes produced with plantar pressure measurements
  Interventions: Other: block 2; Other: with measurements

INTERVENTIONS:
Other: block 1 — shoemaker 1 produces shoes according to standard methods, shoemaker 2 uses plantar pressure measurements
  Arms: group 1; group 2
Other: block 2 — shoemaker 2 produces shoes according to standard methods, shoemaker 1 uses plantar pressure measurements
  Arms: group 3; group 4
Other: standard — patient wears shoes produced with standard method
  Arms: group 1; group 3
Other: with measurements — patient wears shoes produced with plantar pressure measurements
  Arms: group 2; group 4

SUMMARY:
The purpose of this study is determine whether the use of plantar pressure measurements in the production of customized therapeutic footwear for patients with diabetes and a history of foot ulceration results in lower production costs and more pressure relief, compared to the standard production. A secondary objective is to explore if a difference in durability can be observed in pressure reduction and development of (pre-) ulcerative lesions between the shoes produced with and without plantar pressure measurements.

DETAILED DESCRIPTION:
For each patient two pairs of shoes will be produced by two shoemakers, one using plantar pressure measurements and one according current standard production procedures. The patient will wear one of these two pairs of shoes during a period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* diabetes
* neuropathy
* prescription of therapeutic footwear
* diabetic foot ulcer in the last 5 years
* receiving regular preventive foot care
* written informed consent

Exclusion Criteria:

* peripheral arterial disease
* not motivated to wear therapeutic footwear
* active foot ulcer
* recent vascular intervention
* severe mobility impairment
* amputation more proximal than toes, except a single ray amputation is allowed.
* severe visual impairment
* active cancer
* severe cardiac/ pulmonary failure
* severe oedema
* chronic drug abuse
* severe psychiatric illness
* hospital admission at the time of inclusion
* any condition that may interfere with follow-up visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The cost-effectiveness of shoes produced with and without plantar pressure measurements. | approximately 10 weeks (at delivery of the shoes)

SECONDARY OUTCOMES:
Change in plantar pressure after wearing the therapeutic shoes for 3 months. | approximately 22 weeks (at follow-up)
The number of participants with reported and/ or visible new diabetic foot problems, such as ulcera or pre-ulcerative lesions. | approximately 22 weeks (at follow-up)
  The number of diabetic foot problems serves as an additional measure of the quality of the therapeutic shoes produced.
Differences in production techniques, materials and procedures used by the two shoemakers to produce the two pair of shoes. | approximately 10 weeks (at delivery of the shoes)
  Qualitative measure of differences in production process of the shoes produced with or without plantar pressure measurements.
Differences in plantar pressures between the two shoes produced. | approximately 10 weeks (at delivery of the shoes)
The use and usability of the shoes produced, measured with the questionnaire "Monitor Orthopaedic Shoes". | approximately 22 weeks (at follow-up)
Differences in plantar pressures between the two shoes produced. | approximately 22 weeks (at follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas C Schaper, PhD, MD, Principal Investigator — Maastricht University Medical Center; Hans H Savelberg, PhD, Study Director — Maastricht University
Locations (2):
- Netherlands (2):
  - Maastricht University, Maastricht
  - Smeets Loopcomfort, Sittard